CLINICAL TRIAL: NCT06967831
Title: Using iPSC Derived Human Basal Ganglia Neurons From Patients With Leigh Syndrome for Metabolic Studies, Assay Development, and Drug Repurposing.
Brief Title: Drug Repurposing for Mitochondrial Disorders Using iPSCs Derived Neural Cells
Acronym: cureMILS
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: European Union (Other); German Research Foundation (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Markus Schuelke, M.D., Professor of Neuropediatrics, Charite University, Berlin, Germany
Other Study IDs: EA2_131_13
Record Dates: First submitted 2025-04-20; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Leigh Syndrome (Maternally Inherited, MILS); Leigh Syndrome (AR, AD, XR)
Keywords: mitochondrial disease; drug repurposing; Leigh syndrome; iPSC derived neural cells; off-label compassionate use; dopaminergic neurons; neuronal precursor cells; maternal inheritance; autosomal recessive inheritance; autosomal dominant inheritance; X-chromosomal recessive inheritance
MeSH Terms: conditions — Leigh Disease; Mitochondrial Diseases; Multiple Pterygium Syndrome, Autosomal Dominant | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — [1] human induced pluripotent stem cells (hiPSC) generated from fibroblasts or from blood blood cells of patients with Leigh syndrome. [2] DNA samples extracted from white blood cells of patients with Leigh syndrome. [3] RNA samples extracted from white blood cells, from cultured skin fibroblasts and from iPSC-derived neural cells of patients with Leigh syndrome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Leigh Syndrome (Maternally Inherited, MILS): Patients with Leigh syndrome carrying disease-causing mutations in their mtDNA. This subtype of Leigh syndrome is called Maternally Inherited Leigh Syndrome (MILS)
  Interventions: Procedure: skin biopsy; Other: generation of iPSCs; Diagnostic Test: blood drawing; Drug: off-label compassionate drug use
- Leigh Syndrome (AR, AD, XR): Patients with mitochondrial diseases that are caused by mutations in the nuclear DNA, which may be inherited in an autosomal recessive (AR), autosomal dominant (AD), or X-chromosomal recessive (XR) mode of inheritance.
  Interventions: Procedure: skin biopsy; Other: generation of iPSCs; Diagnostic Test: blood drawing; Drug: off-label compassionate drug use

INTERVENTIONS:
Procedure: skin biopsy — Taking a punch skin biopsy of 3 mm diameter under local anesthesia and culturing skin fibroblasts from them.
Other: generation of iPSCs — Using cultured skin fibroblasts of the patients, iPSCs will be generated according to standard procedures.
Diagnostic Test: blood drawing — Drawing blood from a peripheral vein for DNA and RNA isolation. The degree of heteroplasmy (mutation load) for the mtDNA mutation will be determined in the blood DNA.
Drug: off-label compassionate drug use — In case the investigators identify a positive hit during drug repurposing with FDA and EMA approved substances, they will offer it as off-label compassionate use to patients for whom no standard treatment is available.

SUMMARY:
In this project, the investigators are using iPSC lines derived from patients with Leigh syndrome that carry mutations in the mitochondrial (mtDNA) and in the nuclear DNA (nDNA) to reprogram them into neural progenitor cells and into dopaminergic neurons. The researchers are using this experimental system to screen FDA (Food and Drug Administration, USA) and EMA (European Medicines Agency) approved drugs for a positive effect on Leigh patient-derived neuronal cells (drug repurposing) using various biochemical, optic, and morphological outcome measures. Confirmed positive hits may be used for compassionate off-label use in Leigh patients when no standard treatment is available.

DETAILED DESCRIPTION:
Leigh syndrome is a rare severe hereditary neurological disease that typically manifests during early childhood and is characterized by the progressive loss of motor and intellectual skills. A hallmark of the disease is the degeneration of neuronal cells in the brainstem and in the basal ganglia, particularly the dopaminergic neurons therein. The genetic underpinnings of this condition are multifaceted, encompassing mutations in both nuclear genes and in those contained within the mitochondrial DNA (mtDNA). The investigators hypothesize that these mutations share a common principle in their capacity to induce dysfunction of mitochondrial processes and of bioenergetic metabolism. The precise mechanism underlying neuronal death remains to be elucidated as researchers presently lack suitable disease models. Notably, the generation of a mouse model for mtDNA mutations has not been achieved, necessitating the exclusive reliance on patient derived material for research into the pathogenesis of these diseases. Moreover, there are currently no pathogenesis-based treatment approaches that have been demonstrated to improve patients' symptoms. Here, the investigators aim to utilize reprogramming technologies to engineer innovative human-derived disease models for research into Leigh syndrome. To this end, the investigators plan generating induced pluripotent stem cells (iPSCs) from fibroblasts of different Leigh syndrome patients who carry both nuclear (e.g. in SURF1) and mtDNA mutations (e.g. in MT-ATP6). Pluripotent progenitor cells offer a novel approach to better understand the pathogenesis of genetic diseases. In the case of Leigh syndrome, accessible cells, such as skin or blood cells, are almost never clinically affected. However, the nerve cells of the basal ganglia, which cannot be obtained via biopsies, are predominantly affected. The underlying mechanisms by which these dopaminergic neurons are particularly vulnerable to mitochondrial dysfunction and subsequent death remain to be elucidated. The objective of this study is to differentiate these induced pluripotent stem cells (iPSCs) into neural precursor cells (NPCs) and then into a neuronal cell population that is predominant inside the basal ganglia, such as dopaminergic neurons. Subsequently, a detailed analysis of these neurons will be conducted to ascertain mitochondrial and metabolic parameters, with the objective of elucidating neuronal changes associated with mitochondrial disease. Consequently, based on the identified dysfunction, imaging test procedures will be developed that are aimed at high sample throughput. This should enable high-throughput screening of molecule libraries on patient-specific iPSC-based neuronal cells for drug repurposing. The initial phase of the study has identified four potential metrics to be used for the screening of EMA and FDA approved drugs (repurposing): [1] measurement of the mitochondrial membrane potential using fluorophores, [2] measurement of calcium transients using fluorophores and reporter constructs, [3] measurement of the oxygen consumption rate (OCR) and the extracellular acidification rate (ECAR) using a Seahorse flux analyzer, and [4] investigation of the axonal outgrowth and branching patterns of the iPSC-derived neuronal cells by high-content screening. Compounds for which the investigators are able to confirm a positive effect by the above mentioned read-out methods will subsequently be provided to a selected number of patients for off-label compassionate use in cases where no standard treatment is available.

ELIGIBILITY:
Inclusion Criteria: 1. Patient has a disease causing mutation in one of the genes causing Leigh syndrome if mutated, 2. Patient has the characteristic cranial MRI abnormalities of Leigh syndrome

Exclusion Criteria: 1. bleeding disorder that precludes a skin biopsy, 2. retraction of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (male and female) who are affected by Leigh syndrome and carry a pathogenic mutation in a gene known to be associated with Leigh syndrome
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Reduction of the increased mitochondrial membrane potential | 1 year
  The investigators will measure the mitochondrial membrane potential in Leigh patient iPSC-derived neural cells. If the membrane potential can be normalized, a drug will be considered a positive hit. The membrane potential will be determined indirectly by the fluorescence intensity measurement of a membrane potential sensitive dye (TMRM). The patients' fluorescence readings will be compared to the fluorescence readings of neural cells that have been generated from healthy control iPSCs.

SECONDARY OUTCOMES:
Reconstitution of the neural outgrowth pattern | 1 year
  The invesitgators will measure the neural axonal outgrowth and branching pattern in Leigh patient iPSC-derived neural cells using high content screening. If a normal outgrowth and branching pattern can be reconstituted in the patient iPSC-derived neural cells, a drug will be considered a positive hit. Axonal outgrowth and branching will be determined by high throughput parallel microscopy. This will determine the axonal growth velocity and the number of branch points per axon. Patients' data will be compared to healthy control iPSC-derived neural cells.
Measuring calcium transients in iPSC derived neural cells | 1 year
  The investigators will measure calcium transients in Leigh patient iPSC-derived neural cells after electrical stimuation or after chmical stimulation using histamin. This essay will be used for high content screening. If a normal calcium signalling pattern can be reconstituted, a drug will be considered a positive hit. The mitochondrial calcium content will be determined using a fluorescent reporter construct (CEPIA) that is targeted into the mitochondrial matrix. No calibrated absolute measurements are possible. The calcium transients of the patient iPSC-derived neural cells will be compared to those of healthy control iPSC-derived neural cells.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schuelke, MD, Principal Investigator — CHARITE - UNIVERSITAETSMEDIZIN BERLIN
Locations (2):
- Germany (2):
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Charite - Universtaetsmedizin Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared upon reasonable request. A data accession committee will decide on each request.

REFERENCES:
- [Background] Lorenz C, Lesimple P, Bukowiecki R, Zink A, Inak G, Mlody B, Singh M, Semtner M, Mah N, Aure K, Leong M, Zabiegalov O, Lyras EM, Pfiffer V, Fauler B, Eichhorst J, Wiesner B, Huebner N, Priller J, Mielke T, Meierhofer D, Izsvak Z, Meier JC, Bouillaud F, Adjaye J, Schuelke M, Wanker EE, Lombes A, Prigione A. Human iPSC-Derived Neural Progenitors Are an Effective Drug Discovery Model for Neurological mtDNA Disorders. Cell Stem Cell. 2017 May 4;20(5):659-674.e9. doi: 10.1016/j.stem.2016.12.013. Epub 2017 Jan 26. PMID 28132834
- [Background] Henke MT, Zink A, Diecke S, Prigione A, Schuelke M. Generation of two mother-child pairs of iPSCs from maternally inherited Leigh syndrome patients with m.8993 T > G and m.9176 T > G MT-ATP6 mutations. Stem Cell Res. 2023 Mar;67:103030. doi: 10.1016/j.scr.2023.103030. Epub 2023 Jan 17. PMID 36669241
- [Background] Steiner T, Zink A, Henke MT, Cecchetto G, Buenning M, Rossi A, Schuelke M, Prigione A. RNA-based generation of iPSCs from a boy carrying the mutation m.9185 T>C in the mitochondrial gene MT-ATP6 and from his healthy mother. Stem Cell Res. 2022 Oct;64:102920. doi: 10.1016/j.scr.2022.102920. Epub 2022 Sep 15. PMID 36137325
- [Background] Carli S, Levarlet A, Diodato D, Bertini ES, Martinelli D, Malandrini A, Lopergolo D, Gallus GN, Ganetzky RD, La Morgia C, Carelli V, Primiano G, Dominguez-Gonzalez C, Serrano-Lorenzo P, Martin MA, Ardissone A, Lamperti C, Nicoletta V, Klopstock T, Distelmaier F, Zeng L, Buchner B, Mancuso M, Schuelke M, Prigione A, Garone C. Natural History of Patients With Mitochondrial ATPase Deficiency Due to Pathogenic Variants of MT-ATP6 and MT-ATP8. Neurology. 2025 Apr;104(7):e213462. doi: 10.1212/WNL.0000000000213462. Epub 2025 Mar 20. PMID 40112238
- [Background] Diodato D, Schiff M, Cohen BH, Bertini E, Rahman S; Workshop participants. 258th ENMC international workshop Leigh syndrome spectrum: genetic causes, natural history and preparing for clinical trials 25-27 March 2022, Hoofddorp, Amsterdam, The Netherlands. Neuromuscul Disord. 2023 Aug;33(8):700-709. doi: 10.1016/j.nmd.2023.06.002. Epub 2023 Jun 15. No abstract available. PMID 37541860
- [Background] Inak G, Rybak-Wolf A, Lisowski P, Pentimalli TM, Juttner R, Glazar P, Uppal K, Bottani E, Brunetti D, Secker C, Zink A, Meierhofer D, Henke MT, Dey M, Ciptasari U, Mlody B, Hahn T, Berruezo-Llacuna M, Karaiskos N, Di Virgilio M, Mayr JA, Wortmann SB, Priller J, Gotthardt M, Jones DP, Mayatepek E, Stenzel W, Diecke S, Kuhn R, Wanker EE, Rajewsky N, Schuelke M, Prigione A. Defective metabolic programming impairs early neuronal morphogenesis in neural cultures and an organoid model of Leigh syndrome. Nat Commun. 2021 Mar 26;12(1):1929. doi: 10.1038/s41467-021-22117-z. PMID 33771987